CLINICAL TRIAL: NCT01268657
Title: Intervention for Disabling Anxiety in Older Adults Injured by Falls
Brief Title: Intervention for Anxiety After Falls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Nimali Jayasinghe, Assistant Professor of Psychology in Clinical Psychiatry, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23 MH 09244
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Specific Phobia; Anxiety
Keywords: PTSD; Fear of Falling; Older Adults; Injurious Falls; Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Phobia, Specific; Anxiety Disorders | interventions — Educational Status; Relaxation Therapy; Mindfulness-Based Stress Reduction; Cognitive Restructuring; Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitive Behavioral Exposure Therapy (Experimental)
  Interventions: Behavioral: Education; Behavioral: Relaxation Training; Behavioral: Cognitive Restructuring; Behavioral: Behavioral Activation; Behavioral: Exposure

INTERVENTIONS:
Behavioral: Education — Learning about anxiety
  Other Names: Psychoeducation
Behavioral: Relaxation Training — Learning skills to reduce tension
  Other Names: Relaxation; Stress Reduction; Stress Reduction Training
Behavioral: Cognitive Restructuring — Learning skills needed to cope better with distressing thoughts
  Other Names: Cognitive Reframing; Positive self-talk
Behavioral: Behavioral Activation — Learning to initiate healthy activity
  Other Names: Increasing physical activity
Behavioral: Exposure — Coaching in how to confront avoided thoughts, situations, and people)
  Other Names: Imaginal exposure; In vivo exposure

SUMMARY:
The purpose of this study is to determine whether a brief intervention for disabling anxiety is practical to conduct and beneficial for older adults injured by falls.

DETAILED DESCRIPTION:
Falls are the most commonly occurring cause of traumatic injury among older adults. For many, the consequences include reduced mobility, difficulty performing basic self-care, social isolation, deteriorating health, or even death. Most interventions for falls do not address anxiety in the aftermath of falling.

After an initial study assessment, participants will complete 8 home-based sessions of a Cognitive-Behavioral therapy (CBT). The sessions will be led by a study clinician who will cover the 5 intervention components:(a) education (learning about anxiety and the rationale for treatment); (b) relaxation training (learning skills to reduce tension); (c) cognitive restructuring (learning skills needed to cope better with distressing thoughts); (d) behavioral activation (learning to initiate healthy activity); and (e) exposure (coaching in how to confront avoided thoughts, situations, and people).

Participants will also complete assessments following completion of the intervention and 3 months after completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 65 years
* English-speaking
* injured due to fall
* hospitalized
* returned home < or = 3 months
* ambulatory
* full or subsyndromal PTSD or Fear of Falling
* residing in one of the five boroughs of New York City

Exclusion Criteria:

* Inability to understand assessment questions
* Marked cognitive impairment
* Dementia
* Schizophrenia
* Bipolar Disorder
* Depression with psychotic features
* Delusional Disorder
* Substance Use Disorder or Dependence
* Active suicidal ideation, intent, or plan
* Active homicidal ideation, intent or plan
* Aphasia
* Acute or severe medical illness or life expectancy < 6 months
* Initiated psychotropic medications < 6 weeks prior
* Initiated mental health treatment < 6 weeks prior
* Psychosocial factors that would compromise study participation (such as not having a telephone)

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The Clinician Administered PTSD Scale (CAPS) and Survey of Activities and Fear of Falling in the Elderly (SAFE) will be primary outcomes. | At initial assessment, following completion of intervention, and 3 months after completion of intervention

SECONDARY OUTCOMES:
Beck Anxiety Inventory, Beck Depression Inventory, Reintegration to Normal Living, Health Related Quality of Life, and other measures will be included. | At initial assessment, following completion of intervention, and 3 months after completion of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nimali Jayasinghe, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States